CLINICAL TRIAL: NCT06035614
Title: Efficacy and Safety of 308-nm Excimer Lamp Combined With Tacrolimus vs Tacrolimus as Monotherapy in Treating Vitiligo on Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clarteis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 000001112022
Record Dates: First submitted 2022-10-24; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Vitiligo; Pediatric ALL; Dermatologic Disease; Autoimmune Diseases
Keywords: vitiligo; excimer; 308nm
MeSH Terms: conditions — Vitiligo; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Skin Diseases; Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tacrolimus + excimer light (group A) (Active Comparator): group A, will be treated by Tacrolimus 0.1% ointment twice daily and excimer light 308nm twice weekly (exciplex®)
  Interventions: Device: exciplex; Drug: Tacrolimus ointment
- Tacrolimus (group B) (Active Comparator): group B will start on Tacrolimus 0.1% ointment twice daily alone
  Interventions: Drug: Tacrolimus ointment

INTERVENTIONS:
Device: exciplex — exciplex, excimer lamp 308nm produced by clarteis
  Arms: Tacrolimus + excimer light (group A)
Drug: Tacrolimus ointment — tacrolimus monohydrate ointment 0.1% TACRUS

SUMMARY:
Vitiligo is a auto immune that impact 2% of the global population, regardless from the phototype. Even though it affects patients in a physical way through loss of pigmentation, it is also impacting them on a mental/emotional way.11-12 Current treatments offer a symptomatic solution to patients, however the response rate can be low and results can be slow.

Pediatric patients in vitiligo deserves special care as frequently (50%), the disease onset is before 20 years of age and, in 25% of the cases, it starts before the age of 10 years.13 Also, the current treatments for children are limited since it can involve pain and claustrophobia. The combination therapy of the study could offer a painless and easy treatment to follow.

If the combination of those two therapies can fasten and improve the response rate, this could be a good option to treat this condition not only in children, but also for adults patients.

ELIGIBILITY:
Inclusion Criteria:

* vitiligo and surface area involved of less than10% who are being followed in the outpatient dermatology clinics of King Abdullah University Hospital (KAUH)
* 6 weeks wash out period from previous treatments will be employed to eliminate any effect from such treatments

Exclusion Criteria:

* Skin dermatoses with Kobner phenomenon
* Lupus erythematous
* Pacemakers
* Hyper-photosensitivity
* Melanoma and non-melanoma skin cancers
* Drugs with photosensitizer side effect
* Radiotherapy
* Pregnancy (by principle, nno study available)
* Diseases that are contagious by contact

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
repigmentation rate | 1,2,3 and 4 months
  Baseline, photos will be taken and the exact sites involved will be recorded. The clinical improvement measured by the percentage of repigmentation will be assessed and compared between the two mentioned groups at 1,2, 3 and 4 months.

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdullah University Hospital, Ar Ramtha, Jordan

IPD SHARING:
Plan to Share IPD: No